CLINICAL TRIAL: NCT01600209
Title: Exact CRC Screening Test: Stool Sample Collection Study to Support Assay Validation Testing
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Exact Sciences 2011-N
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Colorectal Cancer
Keywords: Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Provide anonymous, clinically characterized specimens for bio-repository for future colorectal cancer-related test development.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Average risk patients: Subjects will be men and women, 50-84 years of age, inclusive, each with a screening colonoscopy resulting in normal findings.

SUMMARY:
The objective of this study is to confirm the sensitivity and specificity of a stool DNA test for detection of colorectal cancer and pre-cancer.

DETAILED DESCRIPTION:
Patients who have recently undergone a colonoscopy that resulted with normal findings will be asked to submit a stool sample (s) (at least 30 days AFTER colonoscopy).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 50-84 years of age, inclusive.
* Subject is at average risk for development of CRC and has undergone a screening colonoscopy with a normal result at least 30 days and no more than 120 days before providing a stool sample for the study. For the purposes of this study, a "normal" colonoscopy result is defined as no polyps of any size detected or removed (including benign, hyperplastic polyps).
* Subject is able to understand the study procedures, and is able to provide signed consent to participate in the study and authorizes release of relevant protected health information through signing a HIPAA consent.
* Subject is able and willing to provide stool samples at least 30 days and no more than 120 days after undergoing a colonoscopy that resulted in normal findings, according to the written instructions provided to them.

Exclusion Criteria:

* Subject has any condition which, in the opinion of the investigator should preclude participation in the study.
* Subject had any findings on recent or any previous colonoscopy including benign, and/or hyperplastic polyps of any size. (Note: Tissue biopsies that result in no histopathology findings are acceptable.)
* Subject has a history or recent diagnosis of CRC or adenoma.
* Subject has a history of aerodigestive tract cancer.
* Subject has had a positive fecal occult blood test or FIT within the previous six (6) months.
* Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease.
* Subject has had overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding)
* Subject has a diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

  * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
  * Greater than or equal to (>=)2 first-degree relatives who have been diagnosed with colon cancer. (Note: first-degree relatives include parents, siblings and offspring).
  * One first-degree relative with CRC diagnosed before the age of 60.
  * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP).
  * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" of "Lynch Syndrome").
  * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are at average risk of developing colorectal cancer at the time of their colonoscopy and the colonoscopy resulted in normal findings.
Sampling Method: Non-Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Exact CRC diagnostic screening test. | 10 months
  The primary endpoints are point estimates of the sensitivity of the diagnostic tests for detection of colorectal neoplasms.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Lidgard, PhD, Study Chair — Chief Scientific Officer
Locations (13):
- United States (13):
  - Desert Sun Clinical Research, Tucson, Arizona
  - Remek Research, Pomona, California
  - Sharp Rees-Stealy, San Diego, California
  - Southern California Medical Gastroenterology Group, Inc, Santa Monica, California
  - Miami Research Associates, Miami, Florida
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Rockford Gastroenterology Associates, LTD., Rockford, Illinois
  - New Orleans Research Institue, Metairie, Louisiana
  - Columbia Medical Practice, Columbia, Maryland
  - Main Line Gastroenterology, Perkasie, Pennsylvania
  - Professional Quality Research, Inc., Austin, Texas
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute, Sandy City, Utah

REFERENCES:
- [Result] Lidgard GP, Domanico MJ, Bruinsma JJ, Light J, Gagrat ZD, Oldham-Haltom RL, Fourrier KD, Allawi H, Yab TC, Taylor WR, Simonson JA, Devens M, Heigh RI, Ahlquist DA, Berger BM. Clinical performance of an automated stool DNA assay for detection of colorectal neoplasia. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1313-8. doi: 10.1016/j.cgh.2013.04.023. Epub 2013 Apr 29. PMID 23639600